CLINICAL TRIAL: NCT02771340
Title: A Phase 1, Open-label, Multicenter Study Evaluating the Safety and Tolerability, Biologic Activity, Pharmacodynamics, and Pharmacokinetics of Single and Repeated Escalating Intravitreal Doses of ICON-1 in Patients With Uveal Melanoma Who Are Planned to Undergo Enucleation or Brachytherapy
Brief Title: Study Evaluating Single and Repeated Intravitreal Doses of ICON-1 in Patients With Uveal Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Iconic Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IT-003
Record Dates: First submitted 2016-05-06; First posted 2016-05-13 (Estimated); Results first posted 2020-09-14 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Uveal Melanoma; Choroid Neoplasm
MeSH Terms: conditions — Uveal Melanoma; Choroid Neoplasms

ARMS (3):
- ICON-1 0.3 mg Singe Dose (Experimental): Patients will receive a single intravitreal dose of ICON-1 0.3 mg
  Interventions: Biological: ICON-1
- ICON-1 0.3 mg Repeat Dosing (Experimental): Patients will receive two intravitreal doses of ICON-1 0.3 mg, one week apart
  Interventions: Biological: ICON-1
- ICON-1 0.6 mg Repeat Dosing (Experimental): Patients will receive two intravitreal doses of ICON-1 0.6 mg, one week apart
  Interventions: Biological: ICON-1

INTERVENTIONS:
Biological: ICON-1 — Intravitreal injection of ICON-1
  Other Names: human Immuno-conjugate 1

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, biological activity, pharmacokinetics and pharmacodynamic activity of single and repeated escalating intravitreal doses of ICON-1 in patients with primary uveal melanoma who are planned to undergo enucleation or brachytherapy of the affected eye.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of any race at least 18 years of age
* Clinical diagnosis of primary uveal melanoma involving the posterior uveal tract in the study eye
* Planned enucleation or brachytherapy of the study eye due to uveal melanoma

Exclusion Criteria:

* Uveal melanoma in the study eye originating in the anterior uveal tract (iris)
* Hereditary or chronic hemorrhagic or coagulopathy conditions (i.e., hemophilia)
* Woman who is pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-05; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Burian, MD, Study Director — Iconic Therapeutics, Inc.
Locations (8):
- United States (8):
  - San Francisco, California
  - Denver, Colorado
  - Leawood, Kansas
  - Boston, Massachusetts
  - Grand Rapids, Michigan
  - Royal Oak, Michigan
  - Portland, Oregon
  - Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CURE OM (Community United for Research and Education of Ocular Melanoma) — http://www.cureom.org
- See also: Ocular Melanoma Foundation (OMF) — http://www.ocularmelanoma.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ICON-1 0.3 mg Singe Dose | ICON-1 0.3 mg Repeat Dosing | ICON-1 0.6 mg Repeat Dosing
Started | 2 | 3 | 5
Completed | 2 | 3 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ICON-1 0.3 mg Singe Dose | ICON-1 0.3 mg Repeat Dosing | ICON-1 0.6 mg Repeat Dosing | Total
Number analyzed (Participants) | 2 | 3 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.5 (0.7) | 64.3 (4.0) | 56.2 (17.2) | 63.9 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1
  Male | 2 | 3 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 3 | 5 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Adverse Events
Time Frame: 30 days (plus or minus 5 days) after surgical procedure
Measure: Count of Participants; unit: Participants
Arm/Group | ICON-1 0.3 mg Singe Dose | ICON-1 0.3 mg Repeat Dosing | ICON-1 0.6 mg Repeat Dosing
Number analyzed (Participants) | 2 | 3 | 5
Participants
  Number of Participants with Adverse Events | 1 | 3 | 5
  Phototoxic Injury/Surgical Complication | 0 | 1 | 0
  Conjunctival Haemorrhage | 0 | 2 | 3
  Conjunctival hyperaemia | 0 | 1 | 0
  Punctate Keratitis | 0 | 1 | 0
  Iridocyclitis | 1 | 0 | 0
  Intraocular Pressure Increased | 1 | 0 | 2

2. Secondary Outcome: Changes in Plasma Levels of ICON-1.
Time Frame: Baseline to 1 day after last dose of ICON-1
Measure: Number; unit: ng/ml-All LLOQ
Arm/Group | ICON-1 0.3 mg Singe Dose | ICON-1 0.3 mg Repeat Dosing | ICON-1 0.6 mg Repeat Dosing
Number analyzed (Participants) | 2 | 3 | 5
ng/ml-All LLOQ | 0 | 0 | 0

3. Secondary Outcome: Change in Best Corrected Visual Acuity (BCVA) From Baseline to End of Study
Description: Best-corrected visual acuity (BCVA) will be measured for each eye, pre treatment prior to dilating eyes, using standard Early Treatment Diabetic Retinopathy Study (ETDRS)-like retro-illuminated charts. BCVA will be recorded as the total letter score in each eye.
Time Frame: Baseline to on or 1 day prior to surgical procedure day
Population: End-of-Study assessments obtained for brachytherapy (placing radioactive material in the eye) patients only.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | ICON-1 0.3 mg Singe Dose | ICON-1 0.3 mg Repeat Dosing | ICON-1 0.6 mg Repeat Dosing
Number analyzed (Participants) | 1 | 1 | 2
Letters | -3 (4.2) | -4.3 (11.8) | -3.6 (6.9)

ADVERSE EVENTS:
Time Frame: During the course of the study and for 30 days last post injection.
Arm/Group | ICON-1 0.3 mg Singe Dose | ICON-1 0.3 mg Repeat Dosing | ICON-1 0.6 mg Repeat Dosing
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/3 | 0/5
Other Adverse Events (participants affected / at risk) | 1/2 | 3/3 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ICON-1 0.3 mg Singe Dose (N=2) | ICON-1 0.3 mg Repeat Dosing (N=3) | ICON-1 0.6 mg Repeat Dosing (N=5)
Phototoxic Injury/Surgical Complication (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ICON-1 0.3 mg Singe Dose (N=2) | ICON-1 0.3 mg Repeat Dosing (N=3) | ICON-1 0.6 mg Repeat Dosing (N=5)
Conjunctival Haemorrhage (Eye disorders) | 0 (0) | 2 (2) | 3 (3)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Punctate Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Intraocular Pressure Increased (Eye disorders) | 1 (1) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-05): https://cdn.clinicaltrials.gov/large-docs/40/NCT02771340/Prot_SAP_000.pdf